CLINICAL TRIAL: NCT02164084
Title: A Phase 1, Single-center, Double-blind, Randomized, Cross-over, Pharmacokinetics, Safety and Tolerability Study of SB204 8% (NVN1000 Gel) and Vehicle Gel
Brief Title: A 2 Period Cross-over Pharmacokinetic Study of SB204 in Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novan, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NI-AC101
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Acne Vulgaris
Keywords: acne
MeSH Terms: conditions — Acne Vulgaris | interventions — berdazimer sodium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SB204 (Experimental): SB204 8% topically twice daily for 4 days and once on Day 5
  Interventions: Drug: SB204
- Vehicle Gel (Placebo Comparator): Vehicle Gel topically twice daily for 4 days and once on Day 5
  Interventions: Drug: Vehicle Gel

INTERVENTIONS:
Drug: SB204 — SB204 Gel with hydrogel
  Other Names: NVN1000
  Arms: SB204
Drug: Vehicle Gel — Vehicle Gel with hydrogel
  Arms: Vehicle Gel

SUMMARY:
This study will identify how much (if any) drug is absorbed from the skin of subjects with acne vulgaris after topical application of SB204.

DETAILED DESCRIPTION:
This is a single-center, double-blind, randomized, 2 period cross-over study to be conducted in 18 subjects (18 years of age and above) each of whom will receive SB204 8% and Vehicle Gel. Subjects who satisfy the entry criteria will be randomized to SB204 8% or Vehicle Gel in a 1:1 ratio for the first treatment period. Study drug will be applied to the face, upper chest, upper back and shoulders (approximately 17% BSA) twice daily on Days 1- 4 approximately 12 hours apart. On Day 5, the study drug will be applied to the same areas only once, in the morning. Pharmacokinetic (PK) profiling will be performed on Day 1 and Day 5. After a wash out period, subjects will be treated with the alternate product and undergo similar treatment and assessments. The primary assessment is the pharmacokinetic profile of nitrate and silicon as markers for systemic exposure to nitric oxide (nitrate) and NVN1000 (silicon) after topical application of SB204 8% to approximately 17% of the total body surface area.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with an acne severity of moderate or severe and a minimum of 20 inflammatory and 20 non-inflammatory lesions on the face, trunk and shoulders
* 18 years of age and older

Exclusion Criteria:

* Any subject with skin disorders of an acute or chronic nature including psoriasis, eczema, tinea versicolor, etc.
* Subjects who smoke or use tobacco products
* Subjects with methemoglobin level greater than 2% at Screening or Baseline by pulse co-oximeter.
* Subjects with a previous history of methemoglobinemia
* Subjects being treated with nitrates or any drug associated with methemoglobinemia
* Subjects with a known history of HIV, hepatitis, or other blood-borne pathogens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-06; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of nitrate and silicon | After single dose and multiple dose (Day 5) application
  Standard PK parameters including area under the curve (AUC) 0-∞, AUC0-t, Cmax, Cmin, and T1/2, for nitrate and silicon. Calculations may be based on actual and/or baseline-subtracted concentrations for nitrate.

SECONDARY OUTCOMES:
Safety | Safety will be assessed throughout the study duration (up to 7 weeks).
  Physical examinations including vital signs, EKGs, and laboratory assessments (serum chemistry, hematology and urinalysis) will be performed at Screening and during the study. Adverse events will be collected throughout the study.

OTHER OUTCOMES:
Tolerability | During both treatment periods, through last day of treatment.
  During the study, cutaneous tolerability assessments will be made at Day 1 and at the end of each treatment period (Day 5). Erythema, dryness, scaling, stinging/burning and itching will be assessed on a four point scale where 0 = none, 1 = mild, 2 = moderate, and 3 = severe.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Sanabria, MD, Principal Investigator — Spaulding Clinical Research LLC
Locations (1):
- Spaulding Clinical Research, LLC, West Bend, Wisconsin, United States